CLINICAL TRIAL: NCT02092675
Title: Endothelial Dysfunction and Frequent Exacerbator Phenotype in Patient With Chronic Obstructive Pulmonary Disease
Brief Title: Endothelial Dysfunction and Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Andrea Vukic Dugac (Other)
Responsible Party: Sponsor-Investigator, Andrea Vukic Dugac, pulmonary disease specialist, Clinical Hospital Centre Zagreb
Organization: Clinical Hospital Centre Zagreb (Other)
Other Study IDs: ED-1971-HR; ED-1971-UHCZ (Other: University Hospital Centre Zagreb)
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Endothelial Dysfunction
Keywords: Chronic obstructive pulmonary disease; frequent exacerbator; endothelial dysfunction; Flow mediated dilatation; Systemic inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- COPD patients - frequent exacerbator: COPD patients with 2 and more exacerbation in one year
- COPD patients - non frequent exacerbator: COPD patients with less than 2 exacerbation during one year
- control group - healthy smokers: healthy smokers, they do not have COPD

SUMMARY:
The purpose of this study is to investigate the role of endothelial dysfunction in chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is one of the leading causes of death in developed countries. Acute exacerbations and cardiovascular diseases are the major causes of morbidity and mortality in COPD patients. According to the frequency of exacerbations, phenotype "frequent exacerbator" is defined and characterised with severe clinical course and was recognised as an increased risk for cardiovascular mortality. Recent studies considered that systemic inflammation plays a key role in the pathogenesis of COPD and endothelial dysfunction is a suspected link between increased cardiovascular mortality and systemic inflammation in COPD patients. Endothelial dysfunction is assessed by determining flow mediated dilatation index (FMD index) or plasma markers. Previous studies have suggested the presence of endothelial dysfunction in COPD patients, as well as the deterioration of endothelial function during exacerbations of COPD. This study will, for the first time, systematically explore endothelial dysfunction in two phenotypically distinct groups of COPD patients with simultaneous assessment of endothelial function flow mediated dilatation index (FMD index) and plasma markers.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients in stable condition ( without exacerbation min 1 months ago)
* Over 40 years
* History of at least 10 py

Exclusion Criteria:

* acute exacerbation of COPD
* active malignancy
* autoimmune disease
* acute myocardial infarction
* diabetes mellitus with late complications
* congestive heart failure
* women of childbearing potential

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with COPD, smokers and former smokers recruited in an ambulatory basis.
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
difference in endothelial dysfunction | 6 months
  Evidence of difference in endothelial dysfunction between COPD frequent exacerbator phenotype group and COPD non frequent exacerbator phenotype group

SECONDARY OUTCOMES:
difference in pulmonary functional tests | 6 months
  Difference in pulmonary functional test between COPD frequent exacerbator phenotype group and COPD non frequent exacerbator phenotype group

OTHER OUTCOMES:
difference in systemic inflammation | 6 months
  Difference in systemic inflammation between COPD frequent exacerbator phenotype group and COPD non frequent exacerbator phenotype group

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vukic Dugac, Principal Investigator — University Hospital Zagreb
Locations (1):
- Univerity Hospital Centre Zagreb, Zagreb, Croatia, Croatia